CLINICAL TRIAL: NCT05484063
Title: Help Optimise and Mobilise Elders (H.O.M.E)
Acronym: HOME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: JurongHealth (Other Government)
Collaborators: Geriatric Education and Research Institute (Other Government); National Healthcare Group, Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GERI1627
Record Dates: First submitted 2022-06-25; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-06

CONDITIONS: Mobility Limitation; Functional Disturbance
Keywords: Elderly; Geriatric; Mobility; Inpatient; Functional Decline; Mobility Intervention; Gait speed; Maximum distance walked; Cost impact; length of stay; Multidisciplinary; Implementation study; 4Ms (Mobility, Mentation, Medication, What Matters); Nursing screen; Group therapy
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: It is a quasi-experimental design study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group will receive a multicomponent, mobility-focused intervention during the course of inpatient admission.
  Interventions: Other: Multicomponent, mobility-focused intervention
- Control (No Intervention): The control group will receive usual care as per current ward practice.

INTERVENTIONS:
Other: Multicomponent, mobility-focused intervention — The intervention group will receive early therapist review (within one working day of admission to HOME unit), to be mobilised at least three times a day. They will also receive additional group exercise therapy sessions, as well as nurse screening for geriatric syndromes. Besides that, they will be screened for 4Ms (Mobility, Mentation, Medication, What Matters) by doctor on admission.
  Arms: Intervention

SUMMARY:
During hospitalisations, older inpatients commonly face issues such as immobility, loss of independence, and functional decline. This leads them down the cascade of dependency with consequent increased risk of adverse outcomes, institutionalisation as well as higher post-acute care costs. The investigators hypothesize that by implementing a mobility intervention in the inpatient setting, patients would be able to maintain their function upon discharge and avoid the cascade of dependency. As such, the investigators aim to do this by implementing and evaluating a mobility intervention, while optimising reversible factors affecting mobility among inpatients admitted to a geriatric unit in Singapore. The investigators will also examine the cost impact of a mobility focused model of care and also adopt the effectiveness-implementation hybrid Type 2 design where both effectiveness and implementation spheres are tested simultaneously.

DETAILED DESCRIPTION:
Aim 1: To examine the effectiveness of multicomponent, mobility-focused model of care in reducing iatrogenic complications and improving patient outcomes. Adopting the Institute for Healthcare Improvement's (IHI) 4Ms framework ("Mobility", "Mentation, "Medication", and "What Matters"), the investigators will examine the effectiveness of timely and individually catered mobility interventions which not only increase mobilization but also optimize factors inhibiting mobility for elderly inpatients. It is hypothesized that the mobility outcomes, such as maximum distance walked and mobilization frequency will be significantly improved for patients who receive the intervention compared to those who receive standard care.

Aim 2: To examine the cost impact of a mobility-focused model of care. The investigators will examine whether the cost of these multicomponent, mobility-focused interventions can be offset from cost savings from early mobilisation benefits, by comparing healthcare utilization costs between-groups. Further to that, a cost effectiveness analysis will be performed should functional effectiveness be observed. For the primary cost impact objective, it is hypothesized that the cost savings arising from reduction in bed days of hospitalization and other medical costs incurred during study period will outweigh the cost of implementing this model of care. In addition, it is also hypothesized that the proposed intervention will be cost-effective through achieving better functional outcomes for patients, with lower costs required.

Aim 3: To evaluate the implementation outcomes of multicomponent, mobility-focused model of care in the process of this intervention. It is hypothesized that this intervention will have good acceptability, feasibility, penetration, implementation costs and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Newly admitted patients to the geriatric service
* Aged 75 years and above
* Mobile with or without the use of a walking aid

Exclusion Criteria:

* Vancomycin-resistant enterococcus (VRE) status
* Requires droplet or airborne precautions
* Critically ill
* Haemodynamically instability
* Requires more than 4-hourly parameters
* Systolic blood pressure <90 mmHg
* Heart rate >100beats/min
* Non-ambulant patients
* With advanced dementia (Functional Assessment Staging Scale [FAST] 7 dementia)
* Fulfills direct admission to another subspecialty unit

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-25 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in maximum distance walked | Upon admission and at the point of discharge (an average of 10 days after inclusion. Analysis will take into account the variability of length of stay)
  The total distance covered by the research participant (in meter)
Mobilisation frequency | Through the duration of admission
  Number of times mobilised. The average mobilisation frequency will be calculated by dividing the sum by the number of admission days.

SECONDARY OUTCOMES:
Change in modified barthel score | Upon admission, at discharge (an average of 10 days after inclusion. Analysis will take into account the variability of length of stay), and one-month post discharge
  The score ranges from 0 to 100 with 0 as the worst outcome
Change in gait speed | Upon admission and at discharge (an average of 10 days after inclusion. Analysis will take into account the variability of length of stay)
  4 meter gait speed test (meter/second)
Inpatient length of stay and discharge location | The duration of admission and upon discharge (an average of 10 days after inclusion. Analysis will take into account the variability of length of stay)
  The duration of admission (days) and the location the respective participant is discharged to
Presence of common iatrogenic complications such as delirium, injurious falls, pressure ulcers, and venous thromboembolisms | At discharge (an average of 10 days after inclusion. Analysis will take into account the variability of length of stay)
  Each of the complication will be measured in nominal scale; 0 denotes the absence of the complication while 1 denotes the presence of the complications. The total number of complications arise will be calculated. The greater the number indicates poorer outcome
Gross amount of patient's bill during index admission, considering subsidy level | At discharge (an average of 10 days after inclusion. Analysis will take into account the variability of length of stay)
  The total gross amount of participant's bill during index admission. The subsidy level will be documented
The intervention related costs for group therapy | At discharge (an average of 10 days after inclusion. Analysis will take into account the variability of length of stay)
  The number of group therapy sessions attended by the participant multiply by the cost for one group therapy session. The subsidy level will be documented.

OTHER OUTCOMES:
Mortality | 1-month follow-up post-discharge
  1 denotes survival while 0 denotes the participant passed away
Readmission | 1-month follow-up post-discharge
  The number of readmission due to the index admission within 30 days post discharged
Healthcare utilisation data and associated costs | 1-month follow-up post-discharge
  Number of visits (associated with index admission) to emergency department, specialist outpatient clinic, general practitioner and the associated costs within 30 days post-discharged
Ambulatory status | 1-month follow-up post-discharge
  Self-reported by the participant. Four options: 0 denotes bed-bound, 1 denotes chair-bound, 2 denotes assisted (furniture cruiser, walking frame, rollator frame, quadstick, single point stick); 4 denotes independent
Fall | 1-month follow-up post-discharge
  0 denotes no fall; 1 denotes fall(s) occured (within 30days post-discharged)
Utilisation of community resources | 1-month follow-up post-discharge
  Self-reported by the participant: Five options: 0 denotes home care; 1 denotes day care; 2 denotes meals on wheels; 3 denotes medical escort service; 4 denotes home personal care

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Tan Dr, Principal Investigator — Ng Teng Fong General Hospital; Lau Lay Khoon Dr, Principal Investigator — Geriatric Education and Research Institute
Locations (2):
- Singapore (2):
  - Ng Teng Fong Hospital, Singapore
  - Geriatrics Education and Research Institute, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Working together with Geriatric Education and Research Institute and National Healthcare Group (Health Services & Outcomes Research).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: During study period.
Access Criteria: Via secure platforms (files to be encrypted with password). For the purposes of data sharing and data analysis.

REFERENCES:
- [Background] Olson EV, Johnson BJ, Thompson LF. The hazards of immobility. 1967. Am J Nurs. 1990 Mar;90(3):43-8. No abstract available. PMID 2178421
- [Background] Hirsch CH, Sommers L, Olsen A, Mullen L, Winograd CH. The natural history of functional morbidity in hospitalized older patients. J Am Geriatr Soc. 1990 Dec;38(12):1296-303. doi: 10.1111/j.1532-5415.1990.tb03451.x. PMID 2123911
- [Background] Mate KS, Berman A, Laderman M, Kabcenell A, Fulmer T. Creating Age-Friendly Health Systems - A vision for better care of older adults. Healthc (Amst). 2018 Mar;6(1):4-6. doi: 10.1016/j.hjdsi.2017.05.005. Epub 2017 Aug 1. PMID 28774720
- [Background] Surkan MJ, Gibson W. Interventions to Mobilize Elderly Patients and Reduce Length of Hospital Stay. Can J Cardiol. 2018 Jul;34(7):881-888. doi: 10.1016/j.cjca.2018.04.033. Epub 2018 May 9. PMID 29960617
- [Background] Smith TO, Sreekanta A, Walkeden S, Penhale B, Hanson S. Interventions for reducing hospital-associated deconditioning: A systematic review and meta-analysis. Arch Gerontol Geriatr. 2020 Sep-Oct;90:104176. doi: 10.1016/j.archger.2020.104176. Epub 2020 Jul 6. PMID 32652367
- [Background] Murray ME, Wells TJ, Callen BL. Hospital resource utilization and functional decline of geriatric patients. Nurs Econ. 2003 May-Jun;21(3):114-9. No abstract available. PMID 12847984
- [Background] Loyd C, Markland AD, Zhang Y, Fowler M, Harper S, Wright NC, Carter CS, Buford TW, Smith CH, Kennedy R, Brown CJ. Prevalence of Hospital-Associated Disability in Older Adults: A Meta-analysis. J Am Med Dir Assoc. 2020 Apr;21(4):455-461.e5. doi: 10.1016/j.jamda.2019.09.015. Epub 2019 Nov 14. PMID 31734122
- [Background] Wu HY, Sahadevan S, Ding YY. Factors associated with functional decline of hospitalised older persons following discharge from an acute geriatric unit. Ann Acad Med Singap. 2006 Jan;35(1):17-23. PMID 16470269
- [Background] Boyd CM, Landefeld CS, Counsell SR, Palmer RM, Fortinsky RH, Kresevic D, Burant C, Covinsky KE. Recovery of activities of daily living in older adults after hospitalization for acute medical illness. J Am Geriatr Soc. 2008 Dec;56(12):2171-9. doi: 10.1111/j.1532-5415.2008.02023.x. PMID 19093915
- [Background] Inouye SK, Bogardus ST Jr, Baker DI, Leo-Summers L, Cooney LM Jr. The Hospital Elder Life Program: a model of care to prevent cognitive and functional decline in older hospitalized patients. Hospital Elder Life Program. J Am Geriatr Soc. 2000 Dec;48(12):1697-706. doi: 10.1111/j.1532-5415.2000.tb03885.x. PMID 11129764
- [Background] Liu B, Moore JE, Almaawiy U, Chan WH, Khan S, Ewusie J, Hamid JS, Straus SE; MOVE ON Collaboration. Outcomes of Mobilisation of Vulnerable Elders in Ontario (MOVE ON): a multisite interrupted time series evaluation of an implementation intervention to increase patient mobilisation. Age Ageing. 2018 Jan 1;47(1):112-119. doi: 10.1093/ageing/afx128. PMID 28985310
- [Background] Hastings SN, Sloane R, Morey MC, Pavon JM, Hoenig H. Assisted early mobility for hospitalized older veterans: preliminary data from the STRIDE program. J Am Geriatr Soc. 2014 Nov;62(11):2180-4. doi: 10.1111/jgs.13095. Epub 2014 Oct 30. PMID 25354909
- [Background] Hastings SN, Choate AL, Mahanna EP, Floegel TA, Allen KD, Van Houtven CH, Wang V. Early Mobility in the Hospital: Lessons Learned from the STRIDE Program. Geriatrics (Basel). 2018 Dec;3(4):61. doi: 10.3390/geriatrics3040061. Epub 2018 Sep 26. PMID 30775370
- [Background] Smart DA, Dermody G, Coronado ME, Wilson M. Mobility Programs for the Hospitalized Older Adult: A Scoping Review. Gerontol Geriatr Med. 2018 Nov 1;4:2333721418808146. doi: 10.1177/2333721418808146. eCollection 2018 Jan-Dec. PMID 30450367
- [Background] Hoyer EH, Friedman M, Lavezza A, Wagner-Kosmakos K, Lewis-Cherry R, Skolnik JL, Byers SP, Atanelov L, Colantuoni E, Brotman DJ, Needham DM. Promoting mobility and reducing length of stay in hospitalized general medicine patients: A quality-improvement project. J Hosp Med. 2016 May;11(5):341-7. doi: 10.1002/jhm.2546. Epub 2016 Feb 5. PMID 26849277
- [Background] Lim SH, Ang SY, Ong HK, Lee TZY, Lee TXL, Luo EZ, Thilarajah S. Promotion of mobility among hospitalised older adults: An exploratory study on perceptions of patients, carers and nurses. Geriatr Nurs. 2020 Sep-Oct;41(5):608-614. doi: 10.1016/j.gerinurse.2020.03.015. Epub 2020 Apr 5. PMID 32268947
- [Background] Chan EY, Samsudin SA, Lim YJ. Older patients' perception of engagement in functional self-care during hospitalization: A qualitative study. Geriatr Nurs. 2020 May-Jun;41(3):297-304. doi: 10.1016/j.gerinurse.2019.11.009. Epub 2019 Nov 29. PMID 31787364
- [Background] Raymond MJ, Jeffs KJ, Winter A, Soh SE, Hunter P, Holland AE. The effects of a high-intensity functional exercise group on clinical outcomes in hospitalised older adults: an assessor-blinded, randomised-controlled trial. Age Ageing. 2017 Mar 1;46(2):208-213. doi: 10.1093/ageing/afw215. PMID 27932360
- [Background] Wallin M, Talvitie U, Cattan M, Karppi SL. Construction of group exercise sessions in geriatric inpatient rehabilitation. Health Commun. 2008;23(3):245-52. doi: 10.1080/10410230802055349. PMID 18569053
- [Background] Renner CIe, Outermans J, Ludwig R, Brendel C, Kwakkel G, Hummelsheim H. Group therapy task training versus individual task training during inpatient stroke rehabilitation: a randomised controlled trial. Clin Rehabil. 2016 Jul;30(7):637-48. doi: 10.1177/0269215515600206. Epub 2015 Aug 27. PMID 26316552
- [Background] Durlak JA, DuPre EP. Implementation matters: a review of research on the influence of implementation on program outcomes and the factors affecting implementation. Am J Community Psychol. 2008 Jun;41(3-4):327-50. doi: 10.1007/s10464-008-9165-0. PMID 18322790
- [Background] Kongkasuwan R, Voraakhom K, Pisolayabutra P, Maneechai P, Boonin J, Kuptniratsaikul V. Creative art therapy to enhance rehabilitation for stroke patients: a randomized controlled trial. Clin Rehabil. 2016 Oct;30(10):1016-1023. doi: 10.1177/0269215515607072. Epub 2015 Sep 22. PMID 26396163
- [Background] Graham ID, Logan J, Harrison MB, Straus SE, Tetroe J, Caswell W, Robinson N. Lost in knowledge translation: time for a map? J Contin Educ Health Prof. 2006 Winter;26(1):13-24. doi: 10.1002/chp.47. PMID 16557505
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Lavis JN, Lomas J, Hamid M, Sewankambo NK. Assessing country-level efforts to link research to action. Bull World Health Organ. 2006 Aug;84(8):620-8. doi: 10.2471/blt.06.030312. PMID 16917649